CLINICAL TRIAL: NCT03242044
Title: Resuscitation of Infants With Congenital Diaphragmatic Hernia With an Intact Umbilical Cord
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-0788
Record Dates: First submitted 2017-07-26; First posted 2017-08-08 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Intervention Model Description: This is a pilot feasibility study that will assess maternal and infant tolerance to the protocols as well as the optimal method for performing an advanced resuscitation with an intact umbilical cord. The investigators have randomly chosen 10 study participant to make this assessment and determine methodologies. For this reason study participants will not be randomized. Pregnant women greater than 18 years of age that consent to the protocol will be enrolled in the study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resuscitation with intact umbilical cord (Experimental): This is a one arm study. Pregnant women greater than 18 years of age with a fetus with left or right sided congenital diaphragmatic hernia of age that consent to the protocol will be enrolled in the study. This is a pilot feasibility study that will assess maternal and infant tolerance to resuscitation with an intact umbilical cord as well as the optimal method for performing an advanced resuscitation with the umbilical cord intact. For this reason patients will not be randomized.
  Interventions: Procedure: Congenital diaphragmatic hernia resuscitation with an intact umbilical cord

INTERVENTIONS:
Procedure: Congenital diaphragmatic hernia resuscitation with an intact umbilical cord — 10 infants with left or right sided congenital diaphragmatic hernia will be intubated and ventilation initiated while still attached to the placental circulation through the umbilical cord. In addition, at the same time, a nasogastric tube will be placed in the stomach to drain entrained air and secretions. After 5 minutes of resuscitation with the umbilical cord intact, the umbilical cord will be cut, infants separated from the placenta and resuscitation performed per routine neonatal resuscitation protocols. Feasibility, the optimal approach and maternal and infant tolerance to the procedure will be assessed as part of the study.

SUMMARY:
Congenital diaphragmatic hernia (CDH) is a severe birth defect, with a prevalence of 1:2000 to 1:3000 live births where a defect in the diaphragm results in, herniation of the abdominal contents into the chest with subsequent compression of the intrathoracic structures and respiratory insufficiency after birth. Respiratory insufficiency is managed with intubation and mechanical ventilation. In addition to managing respiratory insufficiency, intubation prevents entrainment of air into the intestines and further compression of the lungs and heart. Resuscitation of infants with CDH also involves placement of a nasogastric tube (NG) into the stomach for removal of entrained air and secretions. As part of routine resuscitation in infants with CDH intubation and NG tube placement are performed after the delivery personnel separates the baby from the placenta by cutting the umbilical cord. This study will assess the feasibility, maternal and fetal tolerance and the optimal approach to performing these initial steps of resuscitation with an intact umbilical cord. The investigators have randomly chosen 10 maternal and infant with congenital diaphragmatic hernia dyads to demonstrate feasibility as well as determine pitfalls and difficulties and the optimal approach to a complex resuscitation with an intact umbilical cord.

DETAILED DESCRIPTION:
CDH is a severe birth defect, with a prevalence of 1:2000 to 1:3000 live births where a defect in the diaphragm results in, herniation of the abdominal contents into the chest with subsequent compression of the intrathoracic structures. Compression of the intrathoracic structures results in pulmonary and left ventricular (LV) hypoplasia and abnormal development of the pulmonary vasculature in utero. These abnormalities in the development of the heart and lungs in utero, result in persistent pulmonary hypertension of the newborn (PPHN) and respiratory insufficiency after birth. Respiratory insufficiency is managed with intubation and mechanical ventilation. In addition to managing respiratory insufficiency, intubation prevents entrainment of air into the intestines and further compression of the lungs and heart. As part of routine resuscitation in infants with CDH intubation is performed after the delivery personnel separates the baby from the placenta by cutting the umbilical cord. Resuscitation of infants with CDH also involves placement of a nasogastric tube (NG) into the stomach for removal of entrained air and secretions as well as placement of catheters in the umbilical artery and vein for administration of medications (vein) and continuous blood pressure monitoring and sampling of blood (artery). As part of routine practice at our institution, these initial steps of resuscitation are all performed in parallel such that while one team is intubating and initiating ventilation as well as placing the NG tube, another team is placing umbilical lines. This approach has allowed the investigators to obtain arterial blood gas samples in 20 infants with CDH at a median of 4 minutes of life (range 2-9 minutes). When compared to cord blood arterial samples, pCO2 increases by a median of 35mmHg (range 11-77mmHg) from a median cord ABG pCO2 of 55mmHg (range 28-78 mmHg) to 88mmHg (range 65-123 mmHg). In addition to these changes in pCO2 median base deficit changed from -2 ± 0.5350 in the arterial cord blood sample to -7.994 ± 0.8547 in the umbilical arterial blood sample. The resultant respiratory and metabolic acidosis decreased the pH from 7.289 ± 0.01946 in the arterial cord blood sample to 7.036 ± 0.02051 after birth. In addition to the above measures, as part of routine resuscitation, the investigators routinely obtain echocardiographic studies in the first hour of life, to guide pulmonary hypertension management. These studies demonstrate left ventricular (LV) dysfunction and right to left shunting at the ductus arteriosus about 50% of the time. The investigators speculate that the LV dysfunction and increased pulmonary vascular resistance are at least in part due to the acidemia described above. In addition, decreased preload to the LV from right to left shunting at the ductus arteriosus also likely contributes to LV dysfunction. Standard of care for infants with marked abnormalities in gas exchange and LV dysfunction is ECMO rescue early on in the delivery room.

Clamping of the umbilical cord is one of the first interventions that occurs after birth. This separates the infant from the placenta, signifying a landmark period during which the newborn transforms into an independent entity. The transition from a fetus to a neonate at birth represents a critical phase in our life. Early or immediate cord clamping is standard practice where delivery of the fetus is followed by immediate clamping of the umbilical cord (<15 seconds). In 2010, the International Liaison Committee on Resuscitation (ILCOR) recommended that cord clamping could be delayed for at least 1 min. Since then for low risk infants, delayed cord clamping has become routine with the delivering providers delaying clamping of the cord for 1 minute prior to initiating routine newborn care. In these low risk infants there have been many published reports demonstrating benefit with delayed cord clamping. The benefits are primarily attributed to an increase in neonatal blood volume, secondary to placenta-fetal transfusion. More recently the benefits of delayed cord clamping have been demonstrated in higher risk infants. In preterm infants, delayed cord clamping decreased the need for inotropic support after birth, decreased the need for blood transfusions and reduced the incidence of necrotizing enterocolitis and intraventricular hemorrhage. These improvements appear more in line with improvements in cardiac function, which may or may not be associated with an increase in blood volume. More recently, in infants with congenital heart disease delayed cord clamping has been shown to be feasible and decreased the need for packed red blood cell transfusions after birth. Despite the benefits of delayed cord clamping on both the cardiopulmonary transition as well as postnatal outcomes, delayed cord clamping has never been employed in infants with congenital diaphragmatic hernia. This is due to the need for immediate resuscitation after birth and the risk of adverse outcomes by delaying the initiation of postnatal care.

In a recent study doppler ultrasound was used to measure arterial and venous umbilical blood flow during delayed cord clamping in term vaginal deliveries. After birth, the probe was placed in the middle of the umbilical cord and pattern and duration of flow in vein and arteries were evaluated until cord clamping. In 90% of infants, umbilical venous flow was still present at 4 minutes and 36 seconds. In 83% of infants, umbilical arterial flow was still present at 4 minutes and 22 seconds and in 72% of infants bidirectional arterial flow was observed. Bidirectional arterial flow appeared at 45 seconds after birth and persisted for a median duration of 2 minutes and 24 seconds (01:37- 03:52). This study implies that placental gas exchange may remain active for at least 4-5 minutes after birth and suggests that delaying cord clamping for 4-5 minutes while initiating resuscitation may be feasible.

In fetal sheep, the effect of initiation of ventilation with an intact umbilical cord was studied by placing flow probes around the ductus arteriosus, carotid and pulmonary arteries and catheters in the carotid and pulmonary arteries for direct pressure measurements. With clamping of the umbilical cord prior to initiation of ventilation, carotid artery and pulmonary artery pressure increased, carotid artery blood flow increased initially and then decreased and pulmonary artery blood flow and right ventricular output decreased. These changes in carotid and pulmonary pressure and flow were accompanied by a decrease in heart rate. With just 30 seconds of ventilation prior to clamping of the umbilical cord, the fluctuations in heart rate, carotid and pulmonary artery pressure and flow were prevented and the cardiopulmonary transition was much more stable.

The first published report of resuscitation with an intact umbilical cord compared 24 hour hematocrit in premature infants (23 0/7-31 6/7 weeks' GA) randomized to 60 seconds of V (initial continuous positive airway pressure) with addition of positive pressure ventilation if needed - delayed cord clamping (DCC), V-DCC or DCC-only where infants were dried and stimulated by gently rubbing the back if apneic. In this study no differences were seen in the peak hematocrit in the first 24 hours, delivery room interventions, early hemodynamics (cerebral oxygenation by near-infrared spectroscopy, cardiac output and stroke volume by electrical cardiometry, or superior vena cava flow by functional echocardiography), or neonatal outcomes. The onset of breathing was similar between both groups however infants receiving DCC received a greater duration of stimulation than V-DCC. While no benefit was seen with V-DCC, no adverse effects were seen and this study demonstrated the feasibility of resuscitation with the cord intact. In addition the primary outcome measure differed from our question of interest as the infants enrolled in this study were low risk for abnormalities in the cardiopulmonary transition.

In this protocol, the investigators propose initiation of resuscitation during the period of delayed cord clamping in infants with congenital diaphragmatic hernia. This is a feasibility study that will assess tolerance of the participants (pregnant mother and their high-risk infants) to this method of resuscitation as well as the optimal setup and approach to resuscitation. Tolerance to this approach would provide these infants the benefits of delayed cord clamping while allowing for simultaneous resuscitation. The first aim of this study is to assess maternal and fetal tolerance to the procedure and determine the optimal approach to resuscitation. In addition to this the investigators will assess if initiation of resuscitation during the period of delayed cord clamping can stabilize gas exchange and prevent the hypercarbia and acidosis that ensues after birth. Due to the physiologic effects of initiation of ventilation prior to clamping of the umbilical cord the investigators hypothesize that initiation of resuscitation prior to umbilical cord clamping will stabilize the cardiopulmonary transition and will decrease the prevalence of LV dysfunction in this population. The results of this study will lay the foundation for a future multi-center randomized trial and are likely to impact the manner in which newborns with CDH are resuscitated after birth

ELIGIBILITY:
Inclusion Criteria:

• Pregnant women 18 years of age and older with a fetus with the diagnosis of left and right sided congenital diaphragmatic hernia who consent to the protocol.

Exclusion Criteria:

* Patients with Morgagni type defects.
* Infants that have undergone fetal endoscopic tracheal occlusion (FETO)
* Infants with CDH with chromosomal anomalies trisomy 18 and 13
* Infants with bilateral congenital diaphragmatic hernia

Max Age: 5 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Tolerance of resuscitation on infants with congenital diaphragmatic hernia with an intact umbilical cord. | 5 minutes
  10 maternal and infant with left or right sided congenital diaphragmatic hernia dyads will be enrolled in the study and maternal and infant tolerance to resuscitation with an intact umbilical cord determined. Maternal tolerance will be assessed by the incidence of post-partum hemorrhage and uterine atony, infant tolerance determined by capillary blood gas assessments of pH, pCO2 and base deficit and the incidence of bradycardia lasting greater than 1 minute.

SECONDARY OUTCOMES:
Feasibility of resuscitation on infants with congenital diaphragmatic hernia with an intact umbilical cord. | 5 minutes
  10 maternal and infant with left or right sided congenital diaphragmatic hernia dyads will be enrolled in the study and feasibility of performing a complex resuscitation with an intact umbilical cord assessed. Feasibility will be assessed by feedback from resuscitation participants as well as efficiency of the resuscitation when compared to historical controls. As part of feasibility the optimal approach to performing the resuscitation with the umbilical cord intact will be determined.
Evaluation of Infant gas exchange after clamping the umbilical cord | 10 minutes
  10 maternal and infant with left or right sided congenital diaphragmatic hernia dyads will be enrolled in the study and after 5 minutes of resuscitation with an intact umbilical cord, the cord will be cut and the infant separated from the mother. Umbilical venous and arterial catheters will be placed and arterial blood gas drawn to assess arterial pH, pCO2, PaO2 and base deficit.
Left ventricular function after resuscitation with an intact umbilical cord | 20 minutes
  10 maternal and infant with left or right sided congenital diaphragmatic hernia dyads will be enrolled in the study and after 5 minutes of resuscitation with an intact umbilical cord, the cord will be cut and the infant separated from the mother. Following separation from the mother echocardiography will be performed on the infant and left ventricular function measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gien, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Results of the study when completed will be published in a peer review journal

REFERENCES:
- [Result] Torfs CP, Curry CJ, Bateson TF, Honore LH. A population-based study of congenital diaphragmatic hernia. Teratology. 1992 Dec;46(6):555-65. doi: 10.1002/tera.1420460605. PMID 1290156
- [Result] Skari H, Bjornland K, Haugen G, Egeland T, Emblem R. Congenital diaphragmatic hernia: a meta-analysis of mortality factors. J Pediatr Surg. 2000 Aug;35(8):1187-97. doi: 10.1053/jpsu.2000.8725. PMID 10945692
- [Result] Harrison MR, Adzick NS, Nakayama DK, deLorimier AA. Fetal diaphragmatic hernia: pathophysiology, natural history, and outcome. Clin Obstet Gynecol. 1986 Sep;29(3):490-501. No abstract available. PMID 3757331
- [Result] Schwartz SM, Vermilion RP, Hirschl RB. Evaluation of left ventricular mass in children with left-sided congenital diaphragmatic hernia. J Pediatr. 1994 Sep;125(3):447-51. doi: 10.1016/s0022-3476(05)83293-7. PMID 8071756
- [Result] Vogel M, McElhinney DB, Marcus E, Morash D, Jennings RW, Tworetzky W. Significance and outcome of left heart hypoplasia in fetal congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2010 Mar;35(3):310-7. doi: 10.1002/uog.7497. PMID 20143332
- [Result] Taira Y, Yamataka T, Miyazaki E, Puri P. Comparison of the pulmonary vasculature in newborns and stillborns with congenital diaphragmatic hernia. Pediatr Surg Int. 1998 Nov;14(1-2):30-5. doi: 10.1007/s003830050429. PMID 9880691
- [Result] Van Loenhout RB, De Krijger RR, Van de Ven CP, Van der Horst IW, Beurskens LW, Tibboel D, Keijzer R. Postmortem biopsy to obtain lung tissue in congenital diaphragmatic hernia. Neonatology. 2013;103(3):213-7. doi: 10.1159/000345921. Epub 2013 Jan 12. PMID 23328121
- [Result] Reiss I, Schaible T, van den Hout L, Capolupo I, Allegaert K, van Heijst A, Gorett Silva M, Greenough A, Tibboel D; CDH EURO Consortium. Standardized postnatal management of infants with congenital diaphragmatic hernia in Europe: the CDH EURO Consortium consensus. Neonatology. 2010;98(4):354-64. doi: 10.1159/000320622. Epub 2010 Oct 27. PMID 20980772
- [Result] Biban P, Filipovic-Grcic B, Biarent D, Manzoni P; International Liaison Committee on Resuscitation (ILCOR); European Resuscitation Council (ERC); American Heart Association (AHA); American Academy of Pediatrics (AAP). New cardiopulmonary resuscitation guidelines 2010: managing the newly born in delivery room. Early Hum Dev. 2011 Mar;87 Suppl 1:S9-11. doi: 10.1016/j.earlhumdev.2011.01.002. Epub 2011 Jan 19. PMID 21251771
- [Result] Niermeyer S, Velaphi S. Promoting physiologic transition at birth: re-examining resuscitation and the timing of cord clamping. Semin Fetal Neonatal Med. 2013 Dec;18(6):385-92. doi: 10.1016/j.siny.2013.08.008. Epub 2013 Sep 19. PMID 24055300
- [Result] Rabe H, Diaz-Rossello JL, Duley L, Dowswell T. Effect of timing of umbilical cord clamping and other strategies to influence placental transfusion at preterm birth on maternal and infant outcomes. Cochrane Database Syst Rev. 2012 Aug 15;(8):CD003248. doi: 10.1002/14651858.CD003248.pub3. PMID 22895933
- [Result] Committee Opinion No. 684: Delayed Umbilical Cord Clamping After Birth. Obstet Gynecol. 2017 Jan;129(1):1. doi: 10.1097/AOG.0000000000001860. PMID 28002310
- [Result] Baenziger O, Stolkin F, Keel M, von Siebenthal K, Fauchere JC, Das Kundu S, Dietz V, Bucher HU, Wolf M. The influence of the timing of cord clamping on postnatal cerebral oxygenation in preterm neonates: a randomized, controlled trial. Pediatrics. 2007 Mar;119(3):455-9. doi: 10.1542/peds.2006-2725. PMID 17332197
- [Result] Vesoulis ZA, Rhoades J, Muniyandi P, Conner S, Cahill AG, Mathur AM. Delayed cord clamping and inotrope use in preterm infants. J Matern Fetal Neonatal Med. 2018 May;31(10):1327-1334. doi: 10.1080/14767058.2017.1315663. Epub 2017 Apr 20. PMID 28372510
- [Result] Rabe H, Reynolds G, Diaz-Rossello J. A systematic review and meta-analysis of a brief delay in clamping the umbilical cord of preterm infants. Neonatology. 2008;93(2):138-44. doi: 10.1159/000108764. Epub 2007 Sep 21. PMID 17890882
- [Result] Mercer JS, Vohr BR, McGrath MM, Padbury JF, Wallach M, Oh W. Delayed cord clamping in very preterm infants reduces the incidence of intraventricular hemorrhage and late-onset sepsis: a randomized, controlled trial. Pediatrics. 2006 Apr;117(4):1235-42. doi: 10.1542/peds.2005-1706. PMID 16585320
- [Result] Backes CH, Huang H, Cua CL, Garg V, Smith CV, Yin H, Galantowicz M, Bauer JA, Hoffman TM. Early versus delayed umbilical cord clamping in infants with congenital heart disease: a pilot, randomized, controlled trial. J Perinatol. 2015 Oct;35(10):826-31. doi: 10.1038/jp.2015.89. Epub 2015 Jul 30. PMID 26226244
- [Result] Boere I, Roest AA, Wallace E, Ten Harkel AD, Haak MC, Morley CJ, Hooper SB, te Pas AB. Umbilical blood flow patterns directly after birth before delayed cord clamping. Arch Dis Child Fetal Neonatal Ed. 2015 Mar;100(2):F121-5. doi: 10.1136/archdischild-2014-307144. Epub 2014 Nov 11. PMID 25389141
- [Result] Hutchon DJ. Ventilation before Umbilical Cord Clamping Improves Physiological Transition at Birth or "Umbilical Cord Clamping before Ventilation is Established Destabilizes Physiological Transition at Birth". Front Pediatr. 2015 Apr 20;3:29. doi: 10.3389/fped.2015.00029. eCollection 2015. No abstract available. PMID 25941666
- [Result] Bhatt S, Alison BJ, Wallace EM, Crossley KJ, Gill AW, Kluckow M, te Pas AB, Morley CJ, Polglase GR, Hooper SB. Delaying cord clamping until ventilation onset improves cardiovascular function at birth in preterm lambs. J Physiol. 2013 Apr 15;591(8):2113-26. doi: 10.1113/jphysiol.2012.250084. Epub 2013 Feb 11. PMID 23401615
- [Result] Katheria A, Poeltler D, Durham J, Steen J, Rich W, Arnell K, Maldonado M, Cousins L, Finer N. Neonatal Resuscitation with an Intact Cord: A Randomized Clinical Trial. J Pediatr. 2016 Nov;178:75-80.e3. doi: 10.1016/j.jpeds.2016.07.053. Epub 2016 Aug 26. PMID 27574999